CLINICAL TRIAL: NCT03177122
Title: Effect of Myo-Inositol- Based Co-treatment on Oocyte Quality in Women With Polycystic Ovarian Syndrome Undergoing Assisted Reproductive Technology
Brief Title: Myo-Inositol- Based Co-treatment in Women With PCOS Undergoing Assisted Reproductive Technology
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Johnny Awwad, Professor of Obstetrics and Gynecology, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AmericanUBMCMYO
Record Dates: First submitted 2017-05-25; First posted 2017-06-06 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Sterility; Infertility
Keywords: Polycystic Ovary Syndrome; Myo-Inositol; Assisted Reproductive Technology; oocyte performance; pregnancy
MeSH Terms: conditions — Infertility; Polycystic Ovary Syndrome | interventions — Inositol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Myo-Inositol (Experimental): 1g Myo-inositol per day, in combination with alpha- lipoic acid and cysteine, (Celine Tablets; Surveal Pharmaceuticals; Belgium) + 400 ug of Folic acid
  Interventions: Drug: Myo-inositol
- No intervention (No Intervention): Standard care: 400 ug of Folic acid

INTERVENTIONS:
Drug: Myo-inositol — Patients belonging to this group will receive 1 gram of Myo-Inositol, in combination with alpha- lipoic acid and cysteine, (Celine Tablets; Surveal Pharmaceuticals; Belgium) starting 6 weeks prior to stimulation and extending until final oocyte maturation, combined with 400 µg of folic acid supplemented daily.
  Other Names: Celine
  Arms: Myo-Inositol

SUMMARY:
This is a prospective comparative randomized controlled study investigating the effect of Myo-Inositol-based co-treatment on oocyte quality measures in women with PCOS.

DETAILED DESCRIPTION:
Polycystic Ovary Syndrome is the most common cause of chronic anovulation in women. Women with PCOS undergoing IVF are at an increased risk for developing both multiple gestation and ovarian hyperstimulation syndrome (OHSS). Since insulin resistance and hyperinsulinemia have been implicated in the pathophysiology of the disorder, the administration of metformin before or during an IVF cycle has been practiced for years in an attempt to improve follicular parameters necessary for reproductive success. Recently, a growing body of evidence has implicated alternative insulin sensitizing drugs, namely Myo-Inositol, in improving various manifestations of the disorder in this women population. Little has been done to evaluate the effect of Myo-Inositol co-treatment on the reproductive performance of PCOS women undergoing Assisted Reproductive Technologies (ART). In this prospective comparative randomized controlled study, women will be randomized into two groups: Women in the control group will receive folic acid daily. Women in the study group will receive Myo-Inositol, in combination with alpha- lipoic acid and cysteine, per day plus folic acid supplemented daily along with ovarian stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40 years at the time of enrollment.
* Women diagnosed with PCOS according to the Rotterdam criteria indicated by oligoamenorrhea (six or fewer menstrual cycles during a period of 1 year), hyperandrogenism (hirsutism, acne, or alopecia) or hyperandrogenemia (elevated levels of total or free T) and typical features of ovaries on ultrasound scan.
* Planned IVF/ICSI treatment.
* Normal uterine cavity (as assessed by hysteroscopy or HSG).
* Normal hormonal investigation: TSH and PRL.

Exclusion Criteria:

* Azoospermia.
* Other medical conditions causing ovulatory disorders, such as hyperprolactinemia, hypothyroidism, or adrenal hyperplasia.
* Hypersensitivity to Myo-Inositol or its derivatives.

Ages: 18 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Oocyte yield | 1 day from ovum pick up
Maturation rate | 1 day from ovum pick up
Fertilization rate | 16-18 hours post insemination

SECONDARY OUTCOMES:
Blood profile (fasting sugar and insulin levels, Testosterone, Sex Hormone-Binding protein, DHEAs, and Androstenedione) | Prior to and 6 weeks post enrollment
Number of gonadotropin ampules | 1 day from oocyte maturation trigger
Obstetrical outcome (preterm birth) | From 24 to 36 weeks gestation
Obstetrical outcome (low birth weight) | From 24 to 36 weeks gestation
Obstetrical outcome (gestational diabetes) | From 24 to 36 weeks gestation
Obstetrical outcome (preeclampsia) | From 24 to 36 weeks gestation
Obstetrical outcome (admission to neonatal intensive care) | From 24 to 36 weeks gestation
Number of stimulation days | 1 day from oocyte maturation trigger
Embryo quality | 3 to 5 days from ovum pick up
Miscarriage rate | 7 weeks post LMP
Ongoing pregnancy | 20 weeks post LMP
Live birth rate | 24 to 42 weeks gestation

CONTACTS AND LOCATIONS:
Overall Officials: Johnny Awwad, MD, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- American University of Beirut Medical Center, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shukla R, Chadha M, Adya A, Yadav A, Singh N, Chauhan RS, Ahmad A, Tiwari RK. Ongoing Clinical Trials for Polycystic Ovarian Syndrome (PCOS) Afflicted Infertility in Women: A Narrative Review. Rev Recent Clin Trials. 2025;20(2):113-123. doi: 10.2174/0115748871325070241008101355. PMID 39421989